CLINICAL TRIAL: NCT06078345
Title: Brown Adipose Tissue as Nutrient Buffer Through Diet Induced Thermogenesis
Acronym: BANDIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: ETH Zurich (Switzerland) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EKNZ 2023-01544
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Brown Adipose Tissue; Metabolic Disease
Keywords: Diet induced thermogenesis; Cold exposure; Energy Expenditure
MeSH Terms: conditions — Metabolic Diseases | interventions — Carbohydrates; CD36 Antigens; Proteins

STUDY DESIGN:
Intervention Model Description: Prospective interventional trial in healthy volunteers with random sequence of the three study interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAT positive (Experimental): Maximal activated supraclavicular BAT SUVmean >1,5 g/ml-
  Interventions: Other: Carbohydrate; Other: Fat; Other: Protein
- BAT negative (Experimental): Maximal activated supraclavicular BAT SUVmean <1,5 g/ml
  Interventions: Other: Carbohydrate; Other: Fat; Other: Protein

INTERVENTIONS:
Other: Carbohydrate — 400 Kcal glucose (100g oGTT)
Other: Fat — 400 Kcal glucose rapeseed oil.
Other: Protein — 400 Kcal Moltein PURE (111g)

SUMMARY:
To test the hypothesis that active BAT improves metabolic health by buffering postprandial metabolites plasma metabolites and energy expenditure will be compared in volunteers with and without active BAT. Both groups will receive test meals with protein, fat and carbohydrates separately, so that the individual impacts of these macronutrients on diet induced thermogenesis and the buffering function of BAT can be derived. BAT biopsies will be taken before and after the test meals for molecular analysis.

DETAILED DESCRIPTION:
In this prospective interventional study healthy individuals will be screened for presence of active BAT: Maximal BAT activity will be achieved by a mild cold stimulus over 2 hous and quantified by 18F-FDG-PET/CT 30 min after injection of 75 MBq of 18F-FDG.

Individuals with FDG-PET positive BAT will be included as BAT-positive subjects (n=15) and individuals with absence of FDG-positive BAT will be included as BAT-negative subjects (n=15) and then take part in three study visits in random order.

During the study visits participants will consume a standardized isocaloric liquid meal consisting of A) glucose (OGTT) B) fat and C) protein.

Energy expenditure will be measured by indirect calorimetry before as well as hourly after the meal for 5 hours. Blood samples will be taken before and at 30 minute intervals after the meal for 5 hours for analysis of blood glucose, triglycerides, FAAs, representative amino acids, insulin and noradrenaline.

Subjects will undergo ultrasound-guided biopsy of the supraclavicular fat depot in the fasting state and after one of the test meals so that biopsies from 5 individuals in each group after each test meal will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 to 28 kg/m2
* Able to give informed consent as documented by signature

Exclusion Criteria:

* Concomitant medication other than prescription free analgesics (paracetamol and NSAID) and oral contraceptives
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, diabetes mellitus)
* Hyper- or hypothyroidism
* Smoker / habitual tobacco use
* Weight change of >5% within 3 months prior to inclusion
* Hypersensitivity to cold (e.g. Raynaud syndrome)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Enrolment into another study using ionizing radiation within the previous 12 months
* Enrolment into another study including a pharmacological or nutritional intervention
* Pregnancy or lactation
* Lab parameters

  * Serum-Creatinine: above 1.5x upper limit of normal (ULN)
  * Glycated Hemoglobin (HbA1c): above 6.0%
  * Random plasma glucose >11 mM

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
AUC Glucose | 1h before and 5 hours after nutritional intervention
  Area under the curve (AUC) of glucose after the oral glucose load in participants with functional BAT as compared to participants without functional BAT

SECONDARY OUTCOMES:
AUC Branched chain amino acids | 1h before and 5 hours after nutritional intervention
  AUC of BCAAs after protein load in in participants with functional BAT as compared to participants without functional BAT
AUC triglycerides | 1h before and 5 hours after nutritional intervention
  AUC of plasma triglycerides after lipid test meal in participants with functional BAT as compared to participants without functional BAT.
Diet induced thermogenesis | 1h before and 5 hours after nutritional intervention
  Diet-induced thermogenesis: AUC of EE above RMR in response to the respective macronutrient (carbohydrate, protein or fat). Measured by indirect calorimetry. The results for each macronutrient will be compared between the BAT positive and BAT negative participants.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias J Betz, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Dept. of Endocrinology, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No